CLINICAL TRIAL: NCT03832309
Title: Non-Pharmacological Techniques to Reduce the Severity and Frequency of Emergency Reactions After Procedural Sedation and Analgesia in the Emergency Department
Brief Title: Techniques to Reduce the Severity and Frequency of Emergent Reactions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough recruitment.
Sponsor: CHRISTUS Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017196
Record Dates: First submitted 2018-08-02; First posted 2019-02-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The study will be conducted in the emergency department at CHRISTUS Spohn Shoreline hospital is the region's primary acute care center. It houses the Chest Pain, Stroke, and Cancer Centers of CHRISTUS Spohn and is the only level II trauma center in south Texas. It is a major affiliate of Texas A& M medical school, and serves an inner-city population
Who Masked: Participant
Masking Description: During the consent for the study, the physician will do the following depending on which group the patient has been randomized to: Packet 1: The physician will be asked to instruct the patient as empathetically and confidently as possible, that the drug the patient will be given will make them feel not pain, cause them to forget the procedure, and allow them to dream the dream of their choice. The resident will specifically ask the patient what he or she wants to dream about and the resident will then write the patient's answer on the instruction sheet. Packet #2: They physician will be asked to read a written statement about how the drug they will be given will cause analgesia, amnesia, and may cause hallucinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Packet 1: The Physician will be asked to instruct the patient as empathetically and confidently as possible, that the drug the patient will be given will make them feel no pain, cause them to forget the procedure, and allow them to dream the dream of their choice.
  Interventions: Behavioral: Do we speak to them in a way that convinces them to have the dream; Behavioral: Speaking to them as a regualar person
- Control Arm (Other): Half of the participants will receive the sedation medication with the usual conversation while the physician is giving the medication to the patient. The other half of the participants will have a more positive conversation, (which is the study intervention), with the physician while being given the medication. Both group's emergence reactions, if any, will be compared to see if the positive conversation reduced the side effect.
  Interventions: Behavioral: Do we speak to them in a way that convinces them to have the dream; Behavioral: Speaking to them as a regualar person

INTERVENTIONS:
Behavioral: Do we speak to them in a way that convinces them to have the dream — During induction, and depending on what group they are randomized to, the physician will speak to them about having a dream while on the drug
Behavioral: Speaking to them as a regualar person — During induction, if the patient is in group 1, the resident performing procedural sedation will remind the patient about what the patient wanted to dream and ask them to focus on that as the ketamine is being administered. If the patient is in group 2, the resident performing procedural sedation will give no specific instruction to the patient at this point.

SUMMARY:
The objectives of this study are first to determine if the power of suggestion will decrease the frequency and severity of emergence reactions after procedural sedation and analgesia with ketamine in the setting of the emergency department. Second, to determine if people dream about what they were thinking about when they were induced with ketamine.

DETAILED DESCRIPTION:
The proposed research will be single blinded (patient) randomized controlled trial with a retrospective component to test the hypothesis that the power of suggestion will reduce the frequency and severity of emergence reactions, even in the setting of the emergency department.

The study will be conducted in the emergency department at CHRISTU Spohn Shoreline Hospital. CHRISTUS Spohn Shore hospital is the region's primary acute care center. It houses the Chest Pain, Stroke, and Cancer Centers of CHRISTUS Spohn, and the only level II trauma center in south Texas. It is a major teaching affiliate of Texas A&M medical school, and serves an inner-city population.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Required need for procedural sedation and analgesia

Exclusion Criteria:

* Age< 18
* Hypertension
* Raised Intracranial pressure
* Major psychological disorders
* Procedures involving laryngel manipulations
* History of Laryngeal sapsm History of adverse reactions to ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
T-Test | 24 months
  Data gathered from post sedation questionnaire, specifically question 5, will be analyzed by comparing the two means of group one and group two using a student's T test,
STAI-6 | 24 months
  To ensure two groups are similar to each other -demographic data, the pre and post opt sedation VAS scores, and the STAI-6 information.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crapo, DO, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Health, Corpus Christi, Texas, United States